CLINICAL TRIAL: NCT00502853
Title: Pilot Study to Evaluate the Effect of Mabthera in Combination With MTX in the Inhibition of Progression of Synovitis, Bone Marrow Edema, and Erosions Evaluated by Magnetic Resonance Imaging (MRI) in the Hand of Patients With Rheumatoid Arthritis.
Brief Title: A Pilot Study of MabThera (Rituximab) Evaluated by MRI in Patients With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21081
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Methotrexate

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15
Drug: Methotrexate — 10-25mg/week

SUMMARY:
This single arm study will measure the effect of MabThera in combination with methotrexate on the progression of synovitis, the extent of bone marrow edema, and the number of erosions in the wrist and hand of patients with rheumatoid arthritis, using a new MRI technique. Patients will receive MabThera 1000mg i.v. on days 1 and 15, in combination with a stable dosage of 10-25mg/week methotrexate throughout the duration of the study. Further courses of MabThera will be provided to eligible patients. MRI will be performed 1-2 weeks before treatment initiation, and repeated 1 and 6 months after the first MabThera infusion. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* rheumatoid arthritis for >=3 months and <=10 years;
* inadequate response to methotrexate (12.5-25mg/week) for >=3 months;
* evidence of erosive disease and/or clinical synovitis in a signal joint.

Exclusion Criteria:

* autoimmune rheumatic diseases other than RA;
* surgical operations on bones/joints in 12 weeks prior to baseline visit;
* concomitant treatment with biologic agents;
* previous treatment with more than one biologic agent approved for RA, or with cell-depleting therapies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10-25 (Actual); Primary Completion 2010-07-23 (Actual); Study Completion 2010-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Università Degli Studi Di Genova - Dimi; Reumatologia, Genoa, Liguria, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus (+) Methotrexate (MTX): Participants received rituximab 1000 milligrams (mg) intravenously (IV) and methylprednisolone 100 mg IV on Days 1 and 15 and MTX at a stable dose of 10-25 mg per week (mg/week) by mouth or parenterally. Nonresponsive participants (defined as Disease Activity Score Based on 28-Joint Count and C-Reactive Protein [DAS28-CRP] score of greater than [>]2.6) could have received additional infusions of rituximab 1000 mg (2 infusions, 14 days apart) provided a minimum of 24 weeks had passed since the first infusion of the last course of study medication.
Period: Overall Study
Arm/Group | Rituximab Plus (+) Methotrexate (MTX)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received any part of an infusion of study drug.
Groups:
- Rituximab + MTX: Participants received rituximab 1000 mg IV and methylprednisolone 100 mg IV on Days 1 and 15 and MTX at a stable dose of 10-25 mg/week by mouth or parenterally. Nonresponsive participants (defined as DAS28-CRP score of >2.6) could have received additional infusions of rituximab 1000 mg (2 infusions, 14 days apart) provided a minimum of 24 weeks had passed since the first infusion of the last course of study medication.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.42 (15.681)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Synovitis Score
Description: Extension and degree of synovitis in wrist according to RAMRIS score developed by OMERACT. Synovitis is an area in synovial compartment that shows above normal post-gadolinium enhancement of a thickness greater than width of normal synovium. Synovitis is assessed in 3 wrist regions (distal radioulnar joint; radiocarpal joint; intercarpal and carpometacarpal joints) and in each metacarpophalangeal (MCP) joint. 1st carpometacarpal joint and 1st MCP joint are not scored. Score 0 is normal, and 1-3 (mild, moderate, severe) are by thirds of the presumed maximum volume of enhancing tissue in the synovial compartment. Total synovitis score=the sum of the individual scores (3 wrist regions [range 0-9] or 4 MCP joints [range 0-12]) for an overall range of 0-21, where 0=no damage and maximum score [9, 12, or 21]=most severe damage. Change in synovitis = Follow-up synovitis score - baseline score.
Time Frame: Baseline, Week 4, and Week 24
Population: The Safety Population included all participants who received any portion of the rituximab dose and was used for efficacy and safety analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 3.4 (1.58)
  Week 4 | 2.3 (2.75)
  Change at Week 4 | -1.1 (2.38)
  Week 24 | 2.4 (1.74)
  Change at Week 24 | -1.0 (1.73)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline to Week 4; Test type: Superiority or Other; p = 0.1776, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p = 0.1215, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.2246, Random coefficient model; Slope = -0.1606, Standard Error of Mean 0.1231

2. Primary Outcome: OMERACT RAMRIS Bone Edema Score
Description: Extension and degree of bone edema in the wrist according to the RAMRIS score developed by OMERACT. Bone edema is a lesion within the trabecular bone, with ill-defined margins and signal characteristics consistent with increased water content. Each bone (wrists: carpal bones, distal radius, distal ulna, metacarpal bases; MCP joints: metacarpal heads, phalangeal bases) is scored separately. The scale of 0-3 was based on the proportion of bone with edema, as follows: 0=no edema; 1=1 percent (%) to 33% of bone was edematous; 2 = 34%-66% of bone was edematous; and 3= 67%-100% of bone was edematous. Total bone edema score=sum of the individual scores for an overall range of 0-69, where 0=no edema and 69=most severe edema. Change in bone edema = follow-up bone edema score - baseline score.
Time Frame: Baseline, Weeks 4 and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 23.2 (13.56)
  Week 4 | 23.8 (15.68)
  Change at Week 4 | 0.6 (14.52)
  Week 24 | 24.0 (14.66)
  Change at Week 24 | 0.8 (16.77)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline to Week 4; Test type: Superiority or Other; p = 0.8989, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p = 0.8834, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.8841, Random coefficient model; Slope = 0.1357, Standard Error of Mean 0.9051

3. Primary Outcome: OMERACT RAMRIS Erosion Score
Description: MRI bone erosion measures a sharply marginated bone lesion, with correct juxta-articular localization and typical signal characteristics, which is visible in 2 planes with a cortical break seen in at least 1 plane. Each bone (wrists: carpal bones, distal radius, distal ulna, metacarpal bases; MCP joints: metacarpal heads, phalangeal bases) scored separately. Scale is 0-10 based on proportion of eroded bone compared to assessed bone volume (0=no erosion; 1=1%-10% of bone eroded; 2=11%-20%, etc). For long bones, assessed bone volume is from articular surface (or best estimated position if absent) to depth of 1 centimeter (cm); in carpal bones it is the whole bone. Total erosion score=sum of individual scores for an overall range of 0-230, where 0=no erosion and 230=most severe erosion. Change in erosion=Follow-up erosion score - baseline score.
Time Frame: Baseline, Week 4, and Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 7.9 (3.67)
  Week 4 | 8.1 (3.63)
  Change at Week 4 | 0.2 (1.14)
  Week 24 | 9.1 (4.38)
  Change at Week 24 | 1.2 (2.39)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline to Week 4; Test type: Superiority or Other; p = 0.5911, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p = 0.1475, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.1463, Random coefficient model; Slope = 0.1786, Standard Error of Mean 0.1123

4. Secondary Outcome: Ritchie Articular Index Scores
Description: The Ritchie Articular Index is a graded assessment of tenderness in 26 joint regions. The sum of the grades of tenderness (0=not tender, 1=tender, 2=tender and causes wince, and 3 tender, causes wince and effort to withdraw) elicited by applying firm pressure over the joint margin of articular joints (such as shoulders, elbow, wrists, hips). The scores ranged from 0 (no tenderness) to 78 (most severe tenderness).
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 20.7 (8.30)
  Week 4 | 16.9 (9.49)
  Change at Week 4 | -3.8 (6.78)
  Week 12 | 9.5 (6.72)
  Change at Week 12 | -11.2 (6.11)
  Week 24 | 11.7 (9.60)
  Change at Week 24 | -9.0 (6.50)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.1101, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0003, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0018, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0023, Random coefficient model; Slope = -2.0857, Standard Error of Mean 0.4965

5. Primary Outcome: Early Enhancement Rate (REE)
Description: A low cost, low field dedicated extremity MRI unit was used, which is specifically designed for the examination of peripheral joints. In addition to the standard OMERACT-RAMRIS scoring system, additional data were elaborated by using "dynamic" MRI, i.e. Contrast-Enhanced Dynamic MRI (DCE-MRI). This method evaluates the diffusion of the contrast mean in a series of very short sequences thus providing a diffusion curve which is proportionate to the extent of inflammation in the synovial membrane. Numerical parameters used with this method are the slope in the initial phase (rate of early enhancement - REE) and its "steady state" condition (relative enhancement - RE). REE per second during the first 55 seconds was calculated according to the formula REE55 = (S55-S0)/(S0x55)x100%. The REE shows the slope of the curve of contrast uptake tangential to the α angle and is steeper if inflammation is higher.
Time Frame: Baseline, Weeks 4 and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percent per second
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
percent per second
  Baseline | 0.356 (0.2651)
  Week 4 | 0.489 (0.5110)
  Change at Week 4 | 0.150 (0.4106)
  Week 24 | 0.363 (0.2615)
  Change at Week 24 | -0.012 (0.3227)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.3358, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.9158, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.8877, Random coefficient model; Slope = 0.003418, Standard Error of Mean 0.02345

6. Primary Outcome: Relative Enhancement (RE) Score
Description: A low cost, low field dedicated extremity MRI unit was used, which is specifically designed for the examination of peripheral joints. In addition to the standard OMERACT-RAMRIS scoring system, additional data were elaborated by using "dynamic" MRI (DCE-MRI). This method evaluates the diffusion of the contrast mean in a series of very short sequences thus providing a diffusion curve which is proportionate to the extent of inflammation in the synovial membrane. Numerical parameters used with this method are the slope in the initial phase (REE) and its "steady state" condition (RE).
Time Frame: Baseline, Weeks 4 and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
percent
  Baseline | 66.978 (42.3981)
  Week 4 | 57.889 (51.9276)
  Change at Week 4 | -3.812 (34.3034)
  Week 24 | 40.075 (21.6891)
  Change at Week 24 | -34.450 (32.9609)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.7624, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0212, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0712, Random coefficient model; Slope = -4.2681, Standard Error of Mean 2.0529

7. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: The Stanford HAQ-DI is a participant-reported questionnaire specific for rheumatoid arthritis (RA). It consist of 20 items referring to eight component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item within a domain was scored on a 4-point Likert scale from 0 to 3: 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. The highest score reported by the participant for a domain determined the score for that domain. The overall disability index is computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 1.788 (0.6848)
  Week 4 | 1.471 (0.7976)
  Change at Week 4 | -0.316 (0.3687)
  Week 12 | 0.838 (0.6668)
  Change at Week 12 | -0.950 (0.7997)
  Week 24 | 0.888 (0.7008)
  Change at Week 24 | -0.900 (0.6503)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.0240, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0045, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0018, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0019, Random Coefficient Model; Slope = -0.1964, Standard Error of Mean 0.04524

8. Secondary Outcome: Patient's Global Assessment of Pain
Description: The participant's assessment of their current level of pain on a 0 to 100 millimeter (mm) horizontal VAS. The left-hand extreme of the line was described as "no pain" and the right-hand as "unbearable pain". The participant was asked to mark the line corresponding to their current level of pain and the distance from the left edge was recorded.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
mm
  Baseline | 60.6 (22.75)
  Week 4 | 49.0 (31.73)
  Change at Week 4 | -11.6 (20.38)
  Week 12 | 34.7 (16.77)
  Change at Week 12 | -29.9 (28.27)
  Week 24 | 22.7 (16.92)
  Change at Week 24 | -30.7 (23.69)
Statistical Analysis 1: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0074, Random Coefficient Model; Slope = -6.6294, Standard Error of Mean 1.8623
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.1273, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0132, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.1542, Student's t-test

9. Secondary Outcome: DAS28 Score
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. A DAS28 score of less than or equal to (≤) 3.2 = low disease activity, a DAS28 score of >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 5.735 (0.8099)
  Week 4 | 5.261 (1.5552)
  Change at Week 4 | -0.474 (0.9250)
  Week 12 | 4.307 (1.4552)
  Change at Week 12 | -1.587 (0.9743)
  Week 24 | 4.400 (1.4263)
  Change at Week 24 | -1.335 (1.1425)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.1396, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0050, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0050, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0054, Random coefficient model; Slope = -0.2902, Standard Error of Mean 0.07966

10. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR was determined using the Westergren method. ESR measures how fast red blood cells (erythrocytes) fall to the bottom of a fine glass tube that is filled with the participant's blood. The higher the sedimentation rate the greater the inflammation.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
mm/hr
  Baseline | 72.6 (27.56)
  Week 4 | 63.8 (26.63)
  Change at Week 4 | -15.6 (15.61)
  Week 12 | 48.0 (26.12)
  Change at Week 12 | -30.2 (26.47)
  Week 24 | 53.4 (18.34)
  Change at Week 24 | -19.1 (21.25)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.0254, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0384, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0271, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.0124, Random coefficient model; Slope = -4.7586, Standard Error of Mean 1.5278

11. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP measured by milligrams per deciliter (mg/dL). High levels of CRP are indicators of active inflammation.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
mg/dL
  Baseline | 21.630 (24.1805)
  Week 4 | 23.480 (22.7518)
  Change at Week 4 | 1.850 (16.9261)
  Week 12 | 10.929 (12.2432)
  Change at Week 12 | -10.929 (18.1919)
  Week 24 | 23.410 (26.8998)
  Change at Week 24 | 1.780 (36.7504)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.7376, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.1631, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.8816, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.8835, Random coefficient model; Slope = -0.2927, Standard Error of Mean 1.9408

12. Secondary Outcome: Anti-Cyclic Citrullinated Peptide (Anti-CCP) Autoantibodies Count
Description: Anti-CCP autoantibodies count measured by units per milliliter (U/mL). The anti-CCP autoantibodies bind antigenic determinants that contain the unusual amino acid citrulline. The anti-CCP antibody is a highly specific diagnostic test of RA (though with variable sensitivity) and a marker of joint damage with high prognostic significance.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
U/mL
  Baseline | 55.230 (33.3902)
  Week 4 | 44.311 (28.4448)
  Change at Week 4 | -10.133 (18.0815)
  Week 12 | 41.925 (32.2708)
  Change at Week 12 | -12.862 (16.7306)
  Week 24 | 122.230 (247.7763)
  Change at Week 24 | 67.000 (247.0019)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.1312, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0662, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.4133, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.6049, Random coefficient model; Slope = 8.8196, Standard Error of Mean 16.4534

13. Secondary Outcome: Rheumatoid Factor (RF) Immunoglobulin M (IgM) Concentrations
Description: RF IgM concentrations measured by international units per milliliter (IU/mL). RF is an antibody reacting against the fragment, crystallizable (Fc) region of IgG. Quantitative measurements have shown a prognostic value in distinguishing between progressive and non-progressive disease in early RA, a correlation with radiologically determined joint damage, and relation with clinical improvement after disease-modifying anti-rheumatic treatment.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
IU/mL
  Baseline | 570.922 (827.0900)
  Week 4 | 307.300 (337.9550)
  Change at Week 4 | -285.138 (530.8209)
  Week 12 | 241.756 (357.8067)
  Change at Week 12 | -329.167 (499.0426)
  Week 24 | 281.230 (337.6633)
  Change at Week 24 | -267.389 (529.7928)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.1725, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.0832, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.1685, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.1331, Random coefficient model; Slope = -55.4458, Standard Error of Mean 33.5821

14. Secondary Outcome: Total Immunoglobulin (Ig) Concentrations
Description: Total Ig concentrations as measured by milligrams per milliliter (mg/mL).
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
mg/mL
  Baseline | 20.258 (6.7055)
  Week 4 | 17.786 (4.7033)
  Change at Week 4 | -1.602 (3.6846)
  Week 12 | 17.296 (4.1845)
  Change at Week 12 | -2.336 (4.0998)
  Week 24 | 18.354 (4.3432)
  Change at Week 24 | -1.042 (4.5527)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.2938, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.2216, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.5670, Student's t-test

15. Secondary Outcome: Hematocrit Concentration (%)
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
percentage
  Baseline | 36.110 (2.2218)
  Week 4 | 37.860 (1.4315)
  Change at Week 4 | 1.750 (2.9497)
  Week 12 | 37.512 (2.5798)
  Change at Week 12 | 1.350 (4.3065)
  Week 24 | 37.967 (2.6106)
  Change at Week 24 | 1.667 (3.6695)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.0934, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.4047, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.2101, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.1451, Random coefficient model; Slope = 0.3997, Standard Error of Mean 0.2506

16. Secondary Outcome: Percentage of Total B-lymphocytes
Description: Concentration of all B-lymphocytes subtypes was assessed.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
percentage of cells
  Baseline | 24.040 (10.2954)
  Week 4 | 22.430 (8.0601)
  Change at Week 4 | -1.610 (7.1818)
  Week 12 | 30.125 (12.0576)
  Change at Week 12 | 5.562 (11.6748)
  Week 24 | 24.133 (10.2802)
  Change at Week 24 | 1.111 (7.7194)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 4; Test type: Superiority or Other; p = 0.4963, Student's t-test
Statistical Analysis 2: Comparison: Rituximab + MTX; Change from Baseline at Week 12; Test type: Superiority or Other; p = 0.2198, Student's t-test
Statistical Analysis 3: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.6773, Student's t-test
Statistical Analysis 4: Comparison: Rituximab + MTX; Trend over time; Test type: Superiority or Other; p = 0.5531, Random coefficient model; Slope = 0.3688, Standard Error of Mean 0.5987

17. Secondary Outcome: Erosion Score - Right Hand
Description: The erosion score per joint of the hands can range from 0 to 5. Erosions were scored 1 if they were discrete but clearly present, and 2 or 3 if they were larger, depending on the surface area of the joint involved. A score of 3 was given if the erosion was large and extended over the imaginary middle of the bone. A score of 5 was given if a complete collapse of the joint was present or if the full surface of the joint was affected. In each joint, individual erosions were summed up to a maximum of 5. The maximal erosion score for each hand was thus 80, considering the 16 areas for erosions per hand.
Time Frame: Baseline and Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline | 2.50 (2.972)
  Week 24 | 2.19 (2.963)
  Change at Week 24 | -0.44 (1.741)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.5002, Student's t-test

18. Secondary Outcome: Erosion Score - Left Hand
Description: as for outcome 17
Time Frame: Baseline and Week 24
Population: Safety Population; n=number of participants with values for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 10
units on a scale
  Baseline (n=10) | 1.90 (2.558)
  Week 24 (n=8) | 1.75 (2.619)
  Change at Week 24 (n=8) | 0.00 (0.707)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 1.0000, Student's t-test

19. Secondary Outcome: Joint Space Narrowing - Right Hand
Description: Joint space narrowing and joint subluxation or luxation are combined in a single score with a range of 0 to 4. A normal joint space was scored 0. A score of 2 was allowed to a focal narrowing of the joint or to a joint space not sufficiently narrowed to be scored 2. The score of 1 was not to be used when the reader was unsure whether there was joint space narrowing. A generalized narrowing leaving more than 50% of the original joint space present was scored 2. A generalized narrowing leaving less than 50% of the original joint space present was scored 3, and a subluxation of a joint was also scored 3. A bony ankylosis or a complete luxation of the joint was scored 4. A total of 13 joints were evaluated for narrowing and the scores were summed (13 times [x] 4 [maximum per joint]). Each sum was normalized to a scale of 0 (best possible outcome) to 100 (worst possible outcome).
Time Frame: Baseline and Week 24
Population: Safety Population; only participants with values at both Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 8
units on a scale
  Baseline | 10.40 (7.859)
  Week 24 | 10.13 (6.786)
  Change at Week 24 | 0.94 (6.609)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.7002, Student's t-test

20. Secondary Outcome: Joint Space Narrowing - Left Hand
Description: Joint space narrowing and joint subluxation or luxation are combined in a single score with a range of 0 to 4. A normal joint space was scored 0. A score of 2 was allowed to a focal narrowing of the joint or to a joint space not sufficiently narrowed to be scored 2. The score of 1 was not to be used when the reader was unsure whether there was joint space narrowing. A generalized narrowing leaving more than 50% of the original joint space present was scored 2. A generalized narrowing leaving less than 50% of the original joint space present was scored 3, and a subluxation of a joint was also scored 3. A bony ankylosis or a complete luxation of the joint was scored 4. A total of 13 joints were evaluated for narrowing and the scores were summed (13 x 4 [maximum per joint]). Each sum was normalized to a scale of 0 (best possible outcome) to 100 (worst possible outcome).
Time Frame: Baseline and Week 24
Population: Safety Population; only participants with values at both Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rituximab + MTX: Participants received 1000 mg of Rituximab by IV infusion on Days 1 and 15 (considered to be one cycle). Participants also received 10-25 mg/week stable concomitant MTX by mouth or parenterally. Additional cycles of 2 infusions each could be administered provided the following: a minimum of 24 weeks had passed since the first infusion of the last course of study medication; the participant had a DAS28-CRP score of >2.6; the participant had a neutrophil count not below 1.5x10^3/μL; there was an absence of significant cardiac or pulmonary disease, primary or secondary immunodeficiency, and infections.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 8
units on a scale
  Baseline | 8.45 (6.039)
  Week 24 | 9.13 (6.004)
  Change at Week 24 | 2.19 (5.694)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.3132, Student's t-test

21. Secondary Outcome: X-Rays: Right Hand Total Score
Description: Right hand total scores as measured by X-rays examining erosion and joint space narrowing. Total score was calculated as the sum of the erosion score and the joint space narrowing score and scores ranged from 0 (best possible outcome) to 180 (worst possible outcome).
Time Frame: Baseline and Week 24
Population: Safety Population; only participants with values at both Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 8
units on a scale
  Baseline | 12.90 (9.433)
  Week 24 | 12.31 (7.828)
  Change at Week 24 | 0.50 (7.714)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.8597, Student's t-test

22. Secondary Outcome: X-Rays: Left Hand Total Score
Description: Left hand total scores as measured by X-rays examining erosion and joint space narrowing. Total score was calculated as the sum of the erosion score and the joint space narrowing score and ranged from 0 (best possible outcome) to 180 (worst possible outcome).
Time Frame: Baseline and Week 24
Population: Safety Population; only participants with values at both Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 8
units on a scale
  Baseline | 10.35 (7.192)
  Week 24 | 10.88 (6.813)
  Change at Week 24 | 2.19 (6.341)
Statistical Analysis 1: Comparison: Rituximab + MTX; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.3617, Student's t-test

ADVERSE EVENTS:
Time Frame: From baseline up to 24 weeks.
Arm/Group | Rituximab + MTX
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=10)
Atrial fibrillation (Cardiac disorders) | 1
Device related infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=10)
Hypothyroidism (Endocrine disorders) | 1
Apical granuloma (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Urinary tract infection bacterial (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.